CLINICAL TRIAL: NCT06963814
Title: A Safety, Tolerability, Pharmacokinetics, Immunogenicity and Preliminary Efficacy Study of HC006 in Combination With a PD-1 Inhibitor in Patients With Advanced Solid Tumors:A Multicenter, Open-Label, Dose-Escalation and Multiple Cohort Dose Expansion Phase 1b Clinical Trial
Brief Title: Study of HC006 in Combination With a PD-1 Inhibitor in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HC Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BT-HC006-102
Record Dates: First submitted 2025-04-30; First posted 2025-05-09 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HC006+ keytruda Dose Escalation (Experimental)
  Interventions: Drug: HC006; Drug: KEYTRUDA ®( Pembrolizumab)
- HC006 +keytruda Dose Expansion (Experimental)
  Interventions: Drug: HC006; Drug: KEYTRUDA ®( Pembrolizumab)

INTERVENTIONS:
Drug: HC006 — Specified dose on specified days
Drug: KEYTRUDA ®( Pembrolizumab) — Specified dose on specified days

SUMMARY:
This is an open-label, multicenter Phase 1b clinical study to evaluate the safety, tolerability, pharmacokinetics, immunogenicity and preliminary efficacy of HC006 in combination with a PD-1 inhibitor in patients with advanced solid tumors. The trial is divided into two stages: dose-escalation and dose expansion. First, the dose-escalation study is completed to determine the recommended dose for subsequent extension studies, and then the dose expansion study is conducted in the proposed tumors with potential treatment benefits.

DETAILED DESCRIPTION:
HC006 is an IgG1 monoclonal antibody targeting CCR8, which can specifically clear CCR8-positive tumor infiltrating Treg cells without affecting CD8+ T cell function, thus enhancing the anti-tumor immune response. It has a synergistic effect on anti-tumor effects when combined with PD-1 inhibitors. Based on the existing evidence-based medicine, HC006 combined with PD-1 inhibitors is expected to provide additional treatment benefits in addition to PD-1 inhibitors for a variety of malignant solid tumors including colorectal cancer, head and neck squamous cell carcinoma, gastric cancer, non-small cell lung cancer, cervical cancer, breast cancer, esophageal cancer, pancreatic cancer, ovarian cancer, melanoma, urothelial cancer and renal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand this trial and voluntarily sign the informed consent form;
2. Advanced solid tumors diagnosed by histology or cytopathology;
3. Be able to provide archived (within 2 years after the first treatment with study drug) or fresh tumor tissue samples for relevant biological sample analysis required by the protocol;
4. At least one measurable lesion according to RECIST Version 1.1 (patients with only brain lesion as target lesion are not accepted);
5. Eastern United States Oncology Assistance Group (ECOG) performance status score of 0 or 1;
6. The expected survival time is more than 3 months;
7. Adequate organ and bone marrow function
8. Females of childbearing potential must have a negative blood pregnancy test within 7 days prior to the first dose of investigational product and be non-lactating; Eligible patients of childbearing potential (male and female) must agree to use a reliable method of contraception (hormonal or barrier method or abstinence) with their partner for at least 6 months from signing informed consent until after the last dose of study drug. Women of non-childbearing potential may not undergo pregnancy test and contraception (postmenopausal for at least 1 year or surgically sterilized).

Exclusion Criteria:

1. Patients with imaging findings showing tumor invasion of great vessels or unclear demarcation from blood vessels;
2. Patients with combined brain metastasis, meningeal metastasis, spinal cord compression or leptomeningeal disease;
3. Previous treatment with monoclonal antibodies, bispecific antibodies, small molecule compounds and cells targeting CCR8 at any time;
4. Conditions may significantly affect the autoimmune status;
5. Patients with serious, uncontrolled and unrecoverable acute and chronic diseases:
6. Subjects with other malignant tumors within 5 years prior to the first dose of the investigational drug ;
7. Subjects who have undergone major organ surgery (excluding aspiration biopsy) within 4 weeks prior to the first dose of study drug, or have experienced significant trauma, or require elective surgery during the trial;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-07-04 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities(DLTs) | up to 24 months
  Incidence of Dose Limiting Toxicities(DLTs)

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Parameter:Maximum serum concentration (Cmax) | up to 24 months
  Maximum serum concentration (Cmax)
Immunogenicity | up to 24 months
  Incidence of anti-drug antibodies (ADAs) to HC006
Objective Response Rate (ORR) per RECIST 1.1 | up to 24 months
  The sum of the proportions of subjects who achieved CR or PR in imaging evaluation as assessed by the investigator based on RECIST1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided